CLINICAL TRIAL: NCT02282111
Title: EUS-guided Core Needle Biopsy (EUS-CNB) Versus EUS-guided Single-incision With Needle Knife (SINK) for the Diagnosis of Upper Gastrointestinal Subepithelial Lesions - a Multicenter Randomized Controlled Trial
Brief Title: EUS-CNB Versus EUS-SINK for Diagnosis of Upper Gastrointestinal (UGI) Subepithelial Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Equality of results between the two groups at interim analysis
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00028905
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Esophageal Subepithelial Lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS-CNB (Active Comparator): Using a linear EUS with color and pulsed Doppler to scan the area for vessels, the lesion was then sampled with a 22-gauge beveled needle (using the slow capillary suction and fanning techniques with 5 to 15 to-and-fro movements with each pass). A total of 4 passes were performed and after that the procedure terminated.
  Interventions: Device: 22-gauge Procore needle (ProCore, Cook Medical Inc., Winston-Salem, NC)
- SINK (Active Comparator): Using a conventional needle-knife sphincterotome connected to an electrosurgical unit, and under direct endoscopic vision, a 6-12mm linear incision was made from the periphery of the lesion to its highest convexity zone. A conventional biopsy forceps was then deeply introduced through the hole, and 2 bites were obtained per pass. A total of 4 passes were performed by passing the biopsy forceps through the incision on each occasion. The mucosal incision was then closed with endoclips whenever possible.
  Interventions: Device: conventional needle-knife sphincterotome (Microknife XL; Boston Scientific Inc, Natick, Mass)

INTERVENTIONS:
Device: 22-gauge Procore needle (ProCore, Cook Medical Inc., Winston-Salem, NC) — Using a linear EUS with color and pulsed Doppler to scan the area for vessels, the lesion was then sampled with a 22-gauge beveled needle (using the slow capillary suction and fanning techniques with 5 to 15 to-and-fro movements with each pass). A total of 4 passes were performed and after that, the procedure terminated.
  Arms: EUS-CNB
Device: conventional needle-knife sphincterotome (Microknife XL; Boston Scientific Inc, Natick, Mass) — Using a conventional needle-knife sphincterotome connected to an electrosurgical unit, and under direct endoscopic vision, a 6-12mm linear incision was made from the periphery of the lesion to its highest convexity zone. A conventional biopsy forceps was then deeply introduced through the hole, and 2 bites were obtained per pass. A total of 4 passes were performed by passing the biopsy forceps through the incision on each occasion. The mucosal incision was then closed with endoclips whenever possible.
  Arms: SINK

SUMMARY:
This is a single-blinded randomized control trial trying to compare the effectiveness of diagnosis between two techniques employed in tissue sampling for subepithelial tumors (SETs) of the gastrointestinal tract. Over 2 years, patients having SET will be randomized to either get the EUS-guided core needle biopsy (EUS-CNB) or EUS-guided single-incision with needle knife (SINK) technique. This is of grave importance because the diagnosis of the myriad types of SETs is made histologically requiring a good sample.

DETAILED DESCRIPTION:
Upper gastrointestinal (GI) subepithelial tumors (SETs) are tumors arising from subepithelial layers of esophageal, gastric or duodenal wall, mostly from the submucosa and muscular layer. The incidence of SETs on routine endoscopy is 0.36% The differential diagnosis of SETs include, though are not limited to: lipoma, leiomyoma, aberrant pancreas, varices, carcinoid, gastrointestinal stromal tumors (GISTs), and lymphomas . Therefore, a correct diagnosis of these tumors is important to guide subsequent management. These lesions are often not accurately diagnosed on cross-sectional imaging . Endoscopic ultrasound (EUS) aids in narrowing the differential diagnosis of the lesion as it is often able to establish the layer of origin . However, an accurate diagnosis and targeted therapy is not made solely on the morphological features but on histologic type and at times mitotic index. Thus the need for techniques to obtain histology is beneficial in guiding management.

Since standard endoscopy with pinch biopsies of the overlying mucosa often fails to provide an adequate sample for analysis, multiple other modalities to sample the lesion have been utilized: EUS-guided fine needle aspiration (EUS-FNA), EUS-guided core needle biopsy (EUS-CNB), bite-on-bite forceps biopsies, EUS-guided single-incision with needle knife (SINK) and endoscopic resection.

EUS-FNA is now considered to be the usual method of sampling; however, the diagnostic yield is low: 38% to 82% . Moreover, EUS-FNA often provides insufficient specimens which may not allow for immunohistochemistry that is often essential for diagnosis . Thus EUS-CNB has been assessed for the purpose of obtaining a core sample which allows for histological assessment. Published data reveals a diagnostic (though not histologic) yield using EUS-CNB of 75% In 2011, the SINK technique for sampling was presented with a reported diagnostic accuracy of 92.8% [8]. The technique utilizes a conventional needle-knife connected to an electrosurgical unit. A 6 to 12-mm mucosal incision is made over the lesion. Then conventional biopsy forceps are introduced to obtain 3-5 samples. Subsequently, the incision is closed with 2 to 3 endoclips.

The purpose of this study is to prospectively compare the efficacy and safety of EUS-CNB with SINK in patients with upper GI SETs. The investigators hypothesis is that the SINK technique will be superior to the EUS-CNB in obtaining a histological specimen. The results of the study would provide data which may improve the diagnostic ability for SETs. This in turn will guide appropriate surveillance or management (surgical or endoscopic) for patients with these lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for EUS evaluation of upper GI SETs measuring an estimated 15mm or greater in maximal diameter.
* Location of SET: esophagus, stomach, duodenum
* Age >18 years and older
* Patient consent obtained

Exclusion Criteria:

* Endoscopically non bulging lesion
* Upper GI SETs <15 mm in size as measured during study EUS
* Lesions not necessitating tissue acquisition: i.e. lipomas, varices
* Cystic lesion
* Patients < 18 years of age
* Uncorrectable Coagulopathy (INR >1,5, platelets <100,000)
* Patients with stigmata of portal hypertension
* Patients with post-surgical UGI anatomy (Roux-en-Y gastric bypass, esophagectomy etc)
* Uncooperative patients
* Pregnant women (women of childbearing age will undergo urine pregnancy testing, which is routine for all endoscopic procedures)
* Refusal to consent form

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouen Khashab, MD, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were excluded from the study because a predominantly cystic lesion was found; the lack of an appreciable mass at Endoscopic Ultrasound scan (EUS).
Groups:
- EUS-CNB: Endoscopic ultrasound-core needle biopsy technique
  22-gauge Procore needle (ProCore, Cook Medical Inc., Winston-Salem, NC): A core-needle was used to take a biopsy from the subepithelial lesion
- EUS-SINK: Endoscopic ultrasound- single incision needle knife technique
  Conventional needle-knife sphincterotome (Microknife XL; Boston Scientific Inc, Natick, Mass): Needle knife sphincterotome was used to take a biopsy of the subepithelial lesion
Period: Overall Study
Arm/Group | EUS-CNB | EUS-SINK
Started | 26 | 30
Completed | 19 | 22
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- EUS-CNB: Endoscopic ultrasound-core needle biopsy technique
  22-gauge Procore needle (ProCore, Cook Medical Inc., Winston-Salem, NC): A core-needle will be used to take a biopsy from the subepithelial lesion
- EUS-SINK: Endoscopic ultrasound- single incision needle knife technique
  conventional needle-knife sphincterotome (Microknife XL; Boston Scientific Inc, Natick, Mass): Needle knife sphincterotome will be used to take a biopsy of the subepithelial lesion
- Total: Total of all reporting groups
Arm/Group | EUS-CNB | EUS-SINK | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (11.9) | 66.2 (13.4) | 67.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Layer of origin [Number; unit: participants]
  Submucosa | 7 | 9 | 16
  Muscularis propria | 17 | 17 | 34
  Indeterminate | 2 | 4 | 6
Echogenicity [Number; unit: participants] — Tissue echogenicity is the ability of a tissue in reflection or transmission of the ultrasound waves as compared to its surrounding tissues. The higher the echogenicity of the tissue is, the whiter it will appear on the ultrasound screen as compared to its surrounding tissues. On the contrary, the lower the echogenicity of the tissue is, the blacker it will appear on the screen.
  participants
    Hypoechoic | 19 | 22 | 41
    Isoechoic | 5 | 7 | 12
    Hyperechoic | 1 | 1 | 2
    Mixed echogenicity | 1 | 0 | 1
Location of the lesion [Number; unit: participants]
  Esophagus | 1 | 1 | 2
  Gastric fundus | 7 | 9 | 16
  Gastric body | 12 | 12 | 24
  Antrum | 4 | 7 | 11
  Doudenum | 2 | 1 | 3
Calcification [Number; unit: participants]
  Yes | 0 | 4 | 4
  No | 26 | 26 | 52
Greatest diameter of the lesion [Median (Inter-Quartile Range); unit: millimeters] | 23.5 [20 to 39] | 25 [20 to 30] | 24.5 [20 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Diagnostic accuracy is defined as the percentage of true positive and true negative biopsy specimens combined divided by total number of specimens
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of all samples
Arm/Group | EUS-CNB | SINK
Number analyzed (Participants) | 19 | 22
percentage of all samples | 94.7 [74.2 to 99] | 95.5 [77.3 to 99.2]

2. Secondary Outcome: Histological Yield
Description: This will be assessed by the percentage of patients whose samples were adequate for histopathological evaluation
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EUS-CNB | SINK
Number analyzed (Participants) | 26 | 30
percentage of participants | 76.9 [57.9 to 88.9] | 86.6 [70.3 to 94.6]

3. Secondary Outcome: Technical Failure Rate
Description: Percentage of procedures in whom sampling technique failed to take biopsy specimens
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of procedures
Arm/Group | EUS-CNB | SINK
Number analyzed (Participants) | 26 | 30
percentage of procedures | 3.3 [0.5 to 16.6] | 3.8 [0.6 to 18.8]

4. Secondary Outcome: Time of the Procedure
Description: Time from the beginning of the incision or needle insertion, to completion of tissue acquisition by the techniques defined in the protocol.
Time Frame: Tissue sampling procedure, up to 60 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | EUS-CNB | SINK
Number analyzed (Participants) | 26 | 30
minutes | 12 [8 to 20] | 11 [8 to 17]

5. Secondary Outcome: Percent Sample Contribution to Immunohistochemistry Diagnosis
Description: Percentage of all samples from participants in whom biopsy specimen was adequate enough to contribute to immunohistochemistry diagnosis
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of all samples
Arm/Group | EUS-CNB | SINK
Number analyzed (Participants) | 19 | 22
percentage of all samples | 94.7 [75.3 to 99] | 86.4 [66.6 to 95.2]

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated from the start of the procedure up to 1 week after the procedure.
Groups:
- EUS-CNB: Using a linear EUS with color and pulsed Doppler to scan the area for vessels, the lesion was then sampled with a 22-gauge beveled needle (using the slow capillary suction and fanning techniques with 5 to 15 to-and-fro movements with each pass). A total of 4 passes were performed and after that, the procedure terminated.
Arm/Group | EUS-CNB | SINK
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/30
Other Adverse Events (participants affected / at risk) | 2/26 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EUS-CNB (N=26) | SINK (N=30)
Delayed bleeding (Surgical and medical procedures) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02282111/Prot_SAP_000.pdf